CLINICAL TRIAL: NCT03460080
Title: Diagnostic Value of AFP-L3 and PIVKA-II in HCC
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Hanoi Medical University (Other)
Collaborators: Bach Mai Hospital (Other)
Responsible Party: Principal Investigator, Bui My Hanh, Director, Science Research and International Cooperation Unit, Hanoi Medical University
Other Study IDs: HMU16222
Record Dates: First submitted 2018-02-12; First posted 2018-03-09 (Actual); Last update posted 2018-03-09 (Actual); Status verified 2018-03

CONDITIONS: Hepatocellular Carcinoma
Keywords: Hepatocellular carcinoma; AFP-L3; PIVKA-II
MeSH Terms: conditions — Carcinoma, Hepatocellular

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Other
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Hepatocellular carcinoma patients: Serum samples are collected before liver resection.
  Interventions: Diagnostic Test: AFP-L3 and PIVKA-II in HCC
- Hepatic hemangioma patients
  Interventions: Diagnostic Test: AFP-L3 and PIVKA-II in HCC

INTERVENTIONS:
Diagnostic Test: AFP-L3 and PIVKA-II in HCC — Serum samples are tested for tumor markers including PIVKA-II, AFP, AFP-L3% and biochemical tests.
  Imaging: CT or MRI

SUMMARY:
The incidence of Hepatocellular carcinoma (HCC) is increasing worldwide. However, most of HCC cases were at advanced stage when the diagnosis established.Early diagnosis improves the prognosis.The study is intended to evaluate the diagnostic efficiency of alpha-fetoprotein-L3 (AFP-L3) and Protein Induced by Vitamin K Absence or antagonist-II (PIVKA-II). This study is performed at Hanoi Medical University Hospital. Participants including patients with HCC and hepatic hemangioma. All the serum samples are collected before any treatments and will be tested in single center in order to decrease bias. Serum samples were tested for PIVKA-II, AFP, AFP-L3 and biochemical indexes including alanine aminotransferase(ALT),aspartate aminotransferase (AST), gamma-glutamyl transferase, HbsAg, Anti HCV, etc.

DETAILED DESCRIPTION:
Hepatocellular carcinoma (HCC) is the third leading cause of cancer deaths worldwide.Early diagnosis improves the prognosis. Protein induced by vitamin K antagonist-II (PIVKA-II), also known as des-γ-carboxyprothrombin (DCP) or acarboxy prothrombin, is an abnormal form of prothrombin induced by vitamin K absence or antagonist-II. The study is intended to evaluate the diagnostic efficiency of AFP-L3 and PIVKA-II. AFP-L3 and PIVKA-II as an effective tumor marker for hepatocellular carcinoma(HCC). Despite the extensive application of PIVKA-II in some hospitals from Vietnam, the diagnostic efficiency including sensitivity, specificity, positive predictive value and negative predictive value still needs more clinical data to evaluate. The research purposes list as follows：1. Determination of changes in AFP-L3 and PIVKA II for HCC.2. Investigating the diagnostic value of AFP-L3 and PIVKA II for HCC. This study is performed at Hanoi Medical University Hospital. Participants including patients with HCC and hepatic hemangioma. All the serum samples are collected before any treatments and will be tested in single center in order to decrease bias. Serum samples were tested for PIVKA-II, AFP, AFP-L3 and biochemical indexes including alanine aminotransferase(ALT),aspartate aminotransferase (AST), gamma-glutamyl transferase, HbsAg, Anti HCV, etc.The diagnosis of HCC was based on HCC criteria of Ministry of Public Health of Vietnam. All HCC diagnoses were confirmed at the time of analysis. Stages of tumor is evaluated by Barcelana classification. The Student's t-test (or Mann-Whitney test) was used to compare continuous variables, and the chi-square test (or Fisher's exact test) was used for categorical variables. A receiver operator characteristic (ROC) curve was used to assess the performance characteristic of PIVKA-II,AFP,AFP-L3 measurement.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 and 85
* Receiving no treatment before diagnosis
* Establishing Diagnosis according to thecriteria of Ministry of Public Health of Vietnam 2012.

Exclusion Criteria:

* Clinical data missing
* Laboratory tests information missing
* Serum samples doesn't qualified
* Obstructive jaundice patients
* Medical history of taking warfarin

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The participants will be recruited through outpatient clinics and inpatient in Hanoi Medical University Hospital.
Sampling Method: Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2018-01-01 (Actual); Primary Completion 2018-11-01 (Estimated); Study Completion 2018-12-01 (Estimated)

PRIMARY OUTCOMES:
PIVKA-II | Day one
  Using PIVKA-II assay kit (chemiluminescent microparticle immunoassay)

SECONDARY OUTCOMES:
Alpha-Fetoprotein (AFP) | Day one
  Using chemiluminescent microparticle immunoassay to measure AFP levels
Alpha-Fetoprotein-L3% (AFP-L3%) | Day one
  Using µTASWako i30 automated immunoassay analyzer to measure AFP-L3% levels
Alanine Aminotransferase (ALT) | Day one
  Using Abbott Architect automated immunoassay analyzer to measure ALT levels
Aspartate Aminotransferase (AST) | Day one
  Using Abbott Architect automated immunoassay analyzer to measure AST levels
Gamma Glutamyl Transferase (γ-GT) | Day one
  Using Abbott Architect automated immunoassay analyzer to measure γ-GT levels
Hepatitis B virus surface antigen (HBsAg) | Day one
  Using Abbott Architect automated immuno-analyzer to measure HBsAg levels
Antibodies to Hepatitis C virus (Anti HCV) | Day one
  Using Abbott Architect automated immunoassay analyzer to measure Anti HCV levels
Albumin | Day one
  Using Abbott Architect automated immunoassay analyzer to measure Albumin levels
Prothrombin Time (PT) (%) | Day one
  Using Abbott Architect automated immunoassay analyzer to measure PT (%)

CONTACTS AND LOCATIONS:
Locations (1):
- Hanoi Medical University, Hanoi, Vietnam

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code